CLINICAL TRIAL: NCT05062681
Title: Randomized Controlled Trial on the Efficacy of Dexamethasone Versus Methyl Prednisolone in Covid-19 Infected Patients With High Oxygen Flow
Brief Title: RCT on the Efficacy of Dexamethasone Versus Methyl Prednisolone in Covid-19 Infected Patients With High Oxygen Flow
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Osama Zayed Mahmoud Rostom, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Steroids in COVID-19
Record Dates: First submitted 2021-09-24; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Pandemic
Keywords: steroids
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Active Comparator): Patients will receive dexamethasone 8 mg q12hours
  Interventions: Drug: Dexamethasone
- methylprednisolone group (Experimental): Patients will receive 1mg/kg/day in 2 divided doses over 30 minutes
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive dexamethasone 8 mg q12hours
  Arms: Dexamethasone group
Drug: Methylprednisolone — Patients will receive 1mg/kg/day in 2 divided doses over 30 minutes
  Arms: methylprednisolone group

SUMMARY:
This study aims to evaluate the therapeutic activity and side effects of 16 mg/day dexamethasone in comparison to equivalent dose of MP (1mg/kg/day)for the management of COVID-19 infected patients.Moreover, and according to the importance of the IL-6/STAT-3 in triggering the inflammatory cascade and as the miRNAs are considered as prognostic markers, hence, the study aims also to study the impact of the used regimens on these biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age) at time of enrolment
2. Present COVID-19 (infection confirmed by RT-PCR or antigen testing)
3. Postive pressure ventilation (non-invasive or invasive) or need supplemental oxygen with non-rebreather mask
4. Admission to ICU in the last 24 hours

Exclusion Criteria:

* 1- Underlying disease requiring chronic corticosteroids 2- Any dose of dexamethasone during the present hospital stay for COVID-19 for ≥5 days before enrollment 3- Systemic corticosteroids during present hospital stay for conditions other than COVID-19 (e.g. septic shock) 4-Any contraindication for corticosteroid administration 5-Cardiac arrest before ICU admission 6-Pregnancy or breast feeding 7- Immunocompromised patients as cancer (active) patients, patients on chemotherapy or radiotherapy, HIV, and transplant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
28 days in hospital mortality | 28 days
  all patients who will die in 28 days from the start of treatment

SECONDARY OUTCOMES:
WHO clinical progression scale | 10 days
  WHO clinical progression scale
Adverse events related to steroids | 10 days
  incidence of infection or hyperglycemia
Duration of ICU stay | 10 days
  Duration of ICU stay
Duration of high oxygen supplementation | 10 days
  Duration of high oxygen supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed EL-Ayashy, Ass. Professor, Study Director — Ass. Professor of Anesthesia and Intensive Care; Mohamed Farouk Abdelsalam, Consultant, Study Chair — Consultant of Clinical Pharmacy and Clinical Nutrition Al-Galaa Military Medical Complex (GMMC)
Locations (1):
- Eman Osama, Cairo, Egypt

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhang J, Xie B, Hashimoto K. Current status of potential therapeutic candidates for the COVID-19 crisis. Brain Behav Immun. 2020 Jul;87:59-73. doi: 10.1016/j.bbi.2020.04.046. Epub 2020 Apr 22. PMID 32334062
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Background] Meduri GU, Bridges L, Shih MC, Marik PE, Siemieniuk RAC, Kocak M. Prolonged glucocorticoid treatment is associated with improved ARDS outcomes: analysis of individual patients' data from four randomized trials and trial-level meta-analysis of the updated literature. Intensive Care Med. 2016 May;42(5):829-840. doi: 10.1007/s00134-015-4095-4. Epub 2015 Oct 27. PMID 26508525
- [Background] Salton F, Confalonieri P, Meduri GU, Santus P, Harari S, Scala R, Lanini S, Vertui V, Oggionni T, Caminati A, Patruno V, Tamburrini M, Scartabellati A, Parati M, Villani M, Radovanovic D, Tomassetti S, Ravaglia C, Poletti V, Vianello A, Gaccione AT, Guidelli L, Raccanelli R, Lucernoni P, Lacedonia D, Foschino Barbaro MP, Centanni S, Mondoni M, Davi M, Fantin A, Cao X, Torelli L, Zucchetto A, Montico M, Casarin A, Romagnoli M, Gasparini S, Bonifazi M, D'Agaro P, Marcello A, Licastro D, Ruaro B, Volpe MC, Umberger R, Confalonieri M. Prolonged Low-Dose Methylprednisolone in Patients With Severe COVID-19 Pneumonia. Open Forum Infect Dis. 2020 Sep 12;7(10):ofaa421. doi: 10.1093/ofid/ofaa421. eCollection 2020 Oct. PMID 33072814
- [Background] Rana MA, Hashmi M, Qayyum A, Pervaiz R, Saleem M, Munir MF, Ullah Saif MM. Comparison of Efficacy of Dexamethasone and Methylprednisolone in Improving PaO2/FiO2 Ratio Among COVID-19 Patients. Cureus. 2020 Oct 12;12(10):e10918. doi: 10.7759/cureus.10918. PMID 33194485
- [Background] Ranjbar K, Moghadami M, Mirahmadizadeh A, Fallahi MJ, Khaloo V, Shahriarirad R, Erfani A, Khodamoradi Z, Saadi MHG. Correction to: Methylprednisolone or dexamethasone, which one is superior corticosteroid in the treatment of hospitalized COVID-19 patients: a triple-blinded randomized controlled trial. BMC Infect Dis. 2021 May 11;21(1):436. doi: 10.1186/s12879-021-06130-7. No abstract available. PMID 33975548
- [Background] Chen L, Lou J, Bai Y, Wang M. COVID-19 Disease With Positive Fecal and Negative Pharyngeal and Sputum Viral Tests. Am J Gastroenterol. 2020 May;115(5):790. doi: 10.14309/ajg.0000000000000610. No abstract available. PMID 32205644
- [Background] Bartel DP. MicroRNAs: target recognition and regulatory functions. Cell. 2009 Jan 23;136(2):215-33. doi: 10.1016/j.cell.2009.01.002. PMID 19167326
- [Background] Correia CN, Nalpas NC, McLoughlin KE, Browne JA, Gordon SV, MacHugh DE, Shaughnessy RG. Circulating microRNAs as Potential Biomarkers of Infectious Disease. Front Immunol. 2017 Feb 16;8:118. doi: 10.3389/fimmu.2017.00118. eCollection 2017. PMID 28261201
- [Background] Guterres A, de Azeredo Lima CH, Miranda RL, Gadelha MR. What is the potential function of microRNAs as biomarkers and therapeutic targets in COVID-19? Infect Genet Evol. 2020 Nov;85:104417. doi: 10.1016/j.meegid.2020.104417. Epub 2020 Jun 8. PMID 32526370
- [Background] Mirzaei R, Mahdavi F, Badrzadeh F, Hosseini-Fard SR, Heidary M, Jeda AS, Mohammadi T, Roshani M, Yousefimashouf R, Keyvani H, Darvishmotevalli M, Sani MZ, Karampoor S. The emerging role of microRNAs in the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. Int Immunopharmacol. 2021 Jan;90:107204. doi: 10.1016/j.intimp.2020.107204. Epub 2020 Nov 13. PMID 33221169
- [Background] Abedi F, Rezaee R, Hayes AW, Nasiripour S, Karimi G. MicroRNAs and SARS-CoV-2 life cycle, pathogenesis, and mutations: biomarkers or therapeutic agents? Cell Cycle. 2021 Jan;20(2):143-153. doi: 10.1080/15384101.2020.1867792. Epub 2020 Dec 31. PMID 33382348
- [Background] Abu-Izneid T, AlHajri N, Ibrahim AM, Javed MN, Salem KM, Pottoo FH, Kamal MA. Micro-RNAs in the regulation of immune response against SARS CoV-2 and other viral infections. J Adv Res. 2021 May;30:133-145. doi: 10.1016/j.jare.2020.11.013. Epub 2020 Dec 2. PMID 33282419
- [Background] Li C, Hu X, Li L, Li JH. Differential microRNA expression in the peripheral blood from human patients with COVID-19. J Clin Lab Anal. 2020 Oct;34(10):e23590. doi: 10.1002/jcla.23590. Epub 2020 Sep 22. PMID 32960473
- [Background] Han H, Ma Q, Li C, Liu R, Zhao L, Wang W, Zhang P, Liu X, Gao G, Liu F, Jiang Y, Cheng X, Zhu C, Xia Y. Profiling serum cytokines in COVID-19 patients reveals IL-6 and IL-10 are disease severity predictors. Emerg Microbes Infect. 2020 Dec;9(1):1123-1130. doi: 10.1080/22221751.2020.1770129. PMID 32475230
- [Background] Liu T, Zhang J, Yang Y, Ma H, Li Z, Zhang J, Cheng J, Zhang X, Zhao Y, Xia Z, Zhang L, Wu G, Yi J. The role of interleukin-6 in monitoring severe case of coronavirus disease 2019. EMBO Mol Med. 2020 Jul 7;12(7):e12421. doi: 10.15252/emmm.202012421. Epub 2020 Jun 5. PMID 32428990
- [Background] Jafarzadeh A, Nemati M, Jafarzadeh S. Contribution of STAT3 to the pathogenesis of COVID-19. Microb Pathog. 2021 May;154:104836. doi: 10.1016/j.micpath.2021.104836. Epub 2021 Mar 7. PMID 33691172
- [Background] Tomazini BM, Maia IS, Cavalcanti AB, Berwanger O, Rosa RG, Veiga VC, Avezum A, Lopes RD, Bueno FR, Silva MVAO, Baldassare FP, Costa ELV, Moura RAB, Honorato MO, Costa AN, Damiani LP, Lisboa T, Kawano-Dourado L, Zampieri FG, Olivato GB, Righy C, Amendola CP, Roepke RML, Freitas DHM, Forte DN, Freitas FGR, Fernandes CCF, Melro LMG, Junior GFS, Morais DC, Zung S, Machado FR, Azevedo LCP; COALITION COVID-19 Brazil III Investigators. Effect of Dexamethasone on Days Alive and Ventilator-Free in Patients With Moderate or Severe Acute Respiratory Distress Syndrome and COVID-19: The CoDEX Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1307-1316. doi: 10.1001/jama.2020.17021. PMID 32876695